CLINICAL TRIAL: NCT02589301
Title: A Single-center, Open-label, Parallel Study With Single Subcutaneous Injection for Pharmacokinetics and Pharmacodynamics Comparison of Two Pegfilgrastim Formulations in Both Male and Female Healthy Volunteers, Test Formulation is an Injectable Solution Containing 6 mg of Pegfilgrastim, Manufactured by Eurofarma Laboratórios S/A, and Reference Formulation (Neulastim® Injectable Solution Containing 6 mg) Marketed by Produtos Roche Químicos e Farmacêuticos S/A
Brief Title: Pharmacokinetics and Pharmacodynamics Comparison Study Between Two Pegfilgrastim Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EF143
Record Dates: First submitted 2015-10-20; First posted 2015-10-28 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-11

CONDITIONS: Neutropenia; Healthy
MeSH Terms: conditions — Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pegfilgrastim (Experimental): Pegfilgrastim (Hematopoietic Growth Factor) injectable solution 6 mg / 0,6mL in a single subcutaneous application.
  Interventions: Biological: Pegfilgrastim
- Neulastim (pegfilgrastim) (Active Comparator): Neulastim injectable solution 6 mg / 0,6mL in a single subcutaneous application.
  Interventions: Biological: Pegfilgrastim

INTERVENTIONS:
Biological: Pegfilgrastim

SUMMARY:
This study will evaluate the pharmacokinetics (relative bioavailability) and pharmacodynamics, after single subcutaneous application, in healthy volunteers of both sexes, between pegfilgrastim formulation, produced by Eurofarma Laboratorios S/A and Neulastim® (reference formulation), marketed by Produtos Roche Químicos e Farmacêuticos S/A.

In addition to that, a pharmacodynamics comparison will be performed, through change in absolute neutrophil count in leukogram performed in the same time of pharmacokinetics analysis collection and through CD34+ cell count in peripheral blood at timepoints 0:00, 96:00 and 384:00 hours.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index equals to or higher than 18.5 and equals to or less than 29.9 kg/m2.
* The volunteer is in good health conditions and does not have clinically significant diseases, as per medical opinion, according to Medical History, measurements of Blood Pressure, Heart Rate and Temperature, Physical Exam, Electrocardiogram, and complementary Laboratorial Exams.
* Able to understand the study nature and objective, including risks and adverse events and who intends to cooperate with the researcher and act according to the whole study requirements, which is confirmed by the signature in the Informed Consent Form.

Exclusion Criteria:

* The volunteer is known to have hypersensitivity to the study drug product or to chemically-related compounds.
* History or presence of hepatic or gastrointestinal diseases or other condition interfering with drug product absorption, distribution, excretion or metabolism.
* Use of maintenance therapy with any drug product, except for oral contraceptive pills.
* History of hepatic, renal, pulmonary, gastrointestinal, neurological, hematological, psychiatric, cardiologic or allergic disease of any etiology requiring pharmacological treatment or that is considered clinically relevant by the researcher.
* Electrocardiographic findings are not recommended by the researcher for participating in the study.
* Results of complementary laboratorial exams outside the values considered normal according to this protocol rules, unless they are considered non-clinically significant by the researcher.
* Smoking.
* Daily intake of more than 5 cups of tea or coffee.
* History of drug or alcohol abuse.
* Use of regular medication within 2 weeks preceding the beginning of this study or use of any medication one week before starting this study.
* Hospital admission for any reason up to 8 weeks before the start of the first study treatment period.
* Treatment in the last 3 months before starting this study treatment with any drug product known to have a well-defined toxic potential in large organs.
* Participation in any pharmacokinetics study with collection of more than 300 mL of blood or intake of any experimental drug product in the last six months before starting the study treatment.
* Donation or loss of 450 mL or more of blood in the last three months preceding the study or donation of more than 1500 mL of blood in the last 12 months before starting the study treatment.
* Reagent result for urine βHCG exam, performed in female volunteers.
* Positive result in urine test for detection of abuse drugs.
* Result higher than 0.1 mg/L in ethylometer test.
* Any condition preventing participation in the study as per researcher's opinion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of comparative pharmacokinetics of pegfilgrastim in healthy volunteers with parameter peak maximum concentration in plasma (Cmax). | 16 days
  A 90% confidence interval (CI) for the differences in transformed data means of test and comparator drugs, for Cmax. The CI antilog obtained constitutes the 90% CI for the ratio of geometric averages of the parameter:
  (Cmax test / Cmax comparator) Formulations are considered statistically bioequivalent if these intervals are between limits of 80% and 125%.
Evaluation of comparative pharmacokinetics of pegfilgrastim in healthy volunteers with parameter area under recombinant G-CSF concentration curve versus time (AUC 0-t). | 16 days
  A 90% confidence interval (CI) for the differences in transformed data means of test and comparator drugs, for AUC 0-t. The CI antilog obtained constitutes the 90% CI for the ratio of geometric averages of the parameter:
  (AUC0-t test / AUC0-t comparator) Formulations are considered statistically bioequivalent if these intervals are between limits of 80% and 125%.
Evaluation of comparative pharmacodynamics of pegfilgrastim in healthy volunteers with parameters: absolute neutrophil count (ANC) versus time. | 16 days

SECONDARY OUTCOMES:
Evaluation of comparative pharmacodynamics of pegfilgrastim in healthy volunteers with CD34+ count versus time. | 6 days
  CD34+ count until 144 hours

CONTACTS AND LOCATIONS:
Overall Officials: José Pedrazzoli Junior, Principal Investigator — Unidade Integrada de Farmacologia e Gastroenterologia
Locations (1):
- Unidade Integrada de Farmacologia e Gastroenterologia, Bragança Paulista, São Paulo, Brazil